CLINICAL TRIAL: NCT06062017
Title: The Effects of Water and Potassium Supplementation on Cardiovascular and Kidney Function in Young Adults
Brief Title: Potassium, Hydration, Cardiovascular, and Kidney Study (PHACKs)
Acronym: PHACKs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Indiana University (Other)
Responsible Party: Principal Investigator, Austin Robinson, Associate Professor, Auburn University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: #23-381
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure; Hydration; Vascular Disease Risk
Keywords: Racial disparities; Hydration; Blood pressure; Vascular function; Potassium
MeSH Terms: interventions — Water

STUDY DESIGN:
Intervention Model Description: After a two-week habitual consumption run-in participants will be assigned to two weeks of water and potassium supplementation.
Masking Description: No masking, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water and Potassium (Experimental): N=40, 20 males, 20 females. Following the two-week habitual run-in period, this group will receive 2000mg potassium supplementation/day for 14 days. This will be achieved by taking capsules filled with potassium chloride powder.
  Interventions: Dietary Supplement: Water and Potassium supplementation
- Habitual consumption (No Intervention): N=40, 20 males, 20 females. All participants will be monitored after two weeks of habitual water and potassium prior to being assigned into two weeks of water and potassium.

INTERVENTIONS:
Dietary Supplement: Water and Potassium supplementation — All Participants will be given cases of water and instructed to drink at least an extra 1L per day. Additionally, participants will be given 2000 mg of potassium via potassium chloride powder.
  Arms: Water and Potassium

SUMMARY:
Compared with White Adults, Non-Hispanic Black Adults are at an elevated risk of developing cardiovascular disease (CVD) and end stage chronic-kidney disease (CKD), two of the leading causes of death in the United States. Inadequate hydration status is associated with risk factors for both CVD and CKD. Prior data show that Black individuals are less likely to be adequately hydrated when compared with their White counterparts. Further, socioeconomic factors have been shown to influence hydration practices. Inadequate hydration influences certain hormones that regulate blood volume and impact blood pressure, but increasing potassium intake may provide some positive effects on normalizing these hormones and blood pressure. Black adults, in particular, are more likely to consume less potassium, have inadequate hydration, and tend to have higher blood pressure. As such, there is a critical need for effective strategies to address racial disparities in hydration and resultant health consequences; as well as establish the role of socioeconomic factors contributing to hydration. Therefore, the investigators are seeking to test the investigators' central hypothesis that water with a potassium supplement will improve hydration and cardiovascular health in young White adults (n = 20, 10 females, 10 males), and to a greater extent in young Black Adults (n = 20, 10 females, 10 males. The investigators will assess measures of blood pressure, arterial stiffness, and biomarkers in the urine and blood samples prior to and following a 14-day hydration intervention of 1) bottled water and 2) bottled water with potassium supplementation (2000mg potassium/day).

DETAILED DESCRIPTION:
Compared with White adults, Non-Hispanic Black adults are at an elevated risk of developing cardiovascular disease (CVD) and end-stage chronic kidney disease (CKD) two of the leading causes of mortality in the United States (U.S.). Inadequate hydration status is associated with all-cause mortality and several risk factors for CVD and CKD including obesity, insulin resistance, hypertension, and metabolic syndrome. Prior data demonstrate Black American individuals are more likely to be hypohydrated (i.e., inadequately hydrated) when compared with White individuals. One study in emerging adults (18-25 years old) indicates that Black adults are more likely to be hypohydrated compared with White adults when assessed using gold-standard 24-hour urine collections. Socioeconomic factors influence hydration practices. For example, there are well-justified increased perceptions of unsafe tap water among racial and ethnic minorities. Indeed, the recent Flint, Michigan, and Jackson, Mississippi water crises have raised public awareness over these environmental injustices and ways to increase safe drinking water availability and access. However, there remains a critical need for empirical studies on 1) strategies to address racial disparities in hydration and resultant health consequences; and 2) the role socioeconomic factors in contributing to hydration.

Importantly, hypohydration is associated with increased production of arginine vasopressin (AVP), a peptide hormone produced in the hypothalamus that influences body water balance via anti-diuretic effects. Plasma copeptin is an established surrogate marker of circulating AVP concentration. Plasma copeptin is associated with incident type 2 diabetes, metabolic syndrome, the progression of CKD, and CVD. Some, but not all, studies have demonstrated racial differences in circulating AVP/copeptin. Further, prior studies that aimed at increasing water resulted in reductions in copeptin and improvements in cardiometabolic health. For example, in a cohort with high plasma copeptin, increased water intake also reduced fasting plasma glucose. In a cohort of adults with overweight and obesity, increased water or low-calorie beverage intake reduced fasting plasma glucose and contributed to modest weight loss. Lastly, over 90% of adults do not meet recommendations for potassium intake. Importantly, potassium improves blood pressure (BP), particularly in Black adults, who tend to consume less potassium and have higher BP. Yet, there remains a knowledge gap regarding whether hydration intervention(s) inclusive of water (with or without) potassium could attenuate racial disparities in hydration status and circulating AVP/copeptin. Therefore, the investigators are seeking to test the investigators' central hypothesis that water with a potassium supplement (2000mg/day) will improve hydration and cardiovascular health in White adults (n = 20, 10 females, 10 males), and to a greater extent in young Black Adults (n = 20, 10 females, 10 males). The investigators will utilize three complementary specific aims to address the investigators' hypotheses:

Aim 1: Determine whether water with potassium supplementation improves hydration status and reduces circulating copeptin. The investigators hypothesize that water and potassium supplementation will improve hydration and renal biomarkers, including increased urine volume, and reduced urine specific gravity, urine osmolality, and plasma copeptin.

Aim 2: Determine whether water with potassium supplementation improves BP and vascular health. The investigators hypothesize that water and potassium supplementation will reduce resting laboratory BP and ambulatory BP (awake, asleep, and nocturnal BP dipping), and reduce arterial stiffness assessed via pulse wave velocity.

Aim 3: Determine whether socioeconomic factors are associated with hydration perceptions, knowledge, and practices. The investigators hypothesize that area deprivation index (ADI, i.e., more deprivation) will be associated with hydration perceptions (e.g., greater distrust of tap water) and inadequate hydration assessed by self-reported fluid intake and urine-specific gravity.

In summary, a knowledge gap remains in determining the underlying reasons for the consistently reported racial differences in hydration. To restate, the purpose of this study is to determine 1) whether prescribing water with potassium supplementation is efficacious at improving hydration and reducing plasma copeptin in Black and White adults; 2) whether improving hydration with supplemental potassium improves BP and vascular function in young Black and White adults; 3) Another area of innovation in the investigators' proposal is determining whether area deprivation index (ADI, i.e., more deprivation) is associated with and 3a) beliefs and practices around hydration and 3b) hydration status. 4) We also seek to determine whether the intervention leads to greater improvements in Black adults who are more likely to be underhydrated.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-30 years
* Resting blood pressure no higher than 150/90 mmHg
* BMI below 35 kg/m2
* Free of any metabolic disease (e.g., diabetes) kidney disease, pulmonary disorders (e.g., COPD), cardiovascular disease (peripheral vascular, cardiac, or cerebrovascular), no autoimmune diseases, and no history of cancer.

Exclusion Criteria:

* Have any precluding medical conditions (i.e. hemophilia) or medication (Pradaxa, Eliquis, etc.) that prevent participants from giving blood.
* Are currently pregnant or trying to become pregnant.
* take any of the following medications that are contraindicated with potassium supplementation:
* Renin-angiotensin-aldosterone system (RAAS) blockers: Candesartan , Eprosartan, Irbesartan, Losartan, Olmesartan, Telmisartan
* Non -steroidal anti-inflammatory medications: Aspirin, Ibuprofen, Naproxen
* Non-selective beta-blockers: Pindolol, Penbutolol, Oxprenolol, Propranolol, Nadolol, Sotalol, Timolol, Tertatolol
* Calcineurin inhibitors: Cyclosporine
* Heparin (or other blood thinning medications)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Urine specific gravity | Change score from habitual consumption to after the hydration interventions (2 weeks)
  24 urine samples will be aliquoted and assessed for urine specific gravity (unitless)
Urine osmolality | Change score from habitual consumption to after the hydration interventions (2 weeks)
  24 urine samples will be aliquoted and assessed for urine osmolality in mOsm/kg (AI Osmometer 3D3)
Urine flow rate | Change score from habitual consumption to after the hydration interventions (2 weeks)
  24 urine samples will be assessed for urine flow rate based on urine volume and self-reported collection time (ml/min).
Plasma copeptin | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Plasma copeptin concentration (picomoles per liter) from a resting blood draw
24-hour ambulatory blood pressure | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Participants will wear an Oscar2 (with SphygmoCor) ambulatory blood pressure monitor on their upper arm for up to 24-hours preceding their study visit to measure systolic and diastolic blood pressure. The purpose of the ambulatory blood pressure monitoring is to determine blood pressure regulation over an entire day. This blood pressure monitor will be set to automatically take blood pressure every 20 minutes. The monitor records and saves each blood pressure measurement automatically.
Pulse wave velocity | Change score from habitual consumption to after the hydration interventions (2 weeks)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave velocity (PWV meters per second). A high-fidelity transducer is used to obtain the pressure waveform at the carotid pulse. Distances from the carotid artery sampling site to the femoral artery (upper leg instrumented with a thigh cuff for oscillometric sphygmomanometry), and from the carotid artery to the suprasternal notch will be recorded. PWV will be expressed as cm/s.
Pulse wave analysis | Change score from habitual consumption to after the hydration interventions (2 weeks)
  The investigators will use the SphygmoCor XCEL system to assess pulse wave analysis (PWA) The sampling site is the brachial artery (upper alarm instrumented with a cuff for oscillometric sphygmomanometer). PWA will be expressed as a percentage (calculated as augmentation pressure divided by the pulse pressure).
Brachial blood pressure | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Seated rachial blood pressure will be measured triplicate after at least 5 minutes of rest using an oscillometric device (Suntech CT 40)

SECONDARY OUTCOMES:
Kidney blood velocity | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Renal and segmental artery blood velocity will be assessed in the decubitis position using a high-frequency ultrasound probe, typically in the range of 3-5 MHz.Using Spectral Doppler, the peak systolic velocity (PSV) in the renal and segmental arteries will be measured.
Plasma Osmolality | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Researchers will analyze blood samples for osmolarity (AI Osmometer 3D3)
Plasma electrolytes | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Researchers will analyze plasma samples for electrolytes (Na, K, Cl) concentration using the SmartLyte Electrolyte Analyzer. The unit of measure for Na, K, and Cl is millimoles per liter (mmol/L).
Blood glucose | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Researchers will analyze whole blood samples for blood glucose concentration in milligrams per deciliter using Cholestech benchtop analyzer
Objective sleep duration | Pre-intervention (14 days)
  Philips actiwatch spectrum will be used to quantify sleep duration in hours. Participants will wear the watch units for 14 days. The investigators will assess sleep duration and cross-check actigraphy wear times with a sleep diary.
Objective sleep efficiency | Pre-intervention (14 days)
  Philips actiwatch spectrum will be used to quantify the percentage of time in bed actually spent sleeping to calculate sleep efficiency.
Subjective sleep duration | Change score from habitual consumption to after the hydration interventions (2 weeks)
  The investigators will use the Pittsburgh Sleep Quality Index (PSQI) to assess sleep duration reflective of the one-month period leading into the study. The global PSQI score can range from 0 to 21 points, however, this outcome specifically refers to self-reported sleep duration in hours.
Subjective sleep quality | Change score from habitual consumption to after the hydration interventions (2 weeks)
  The investigators will use the Pittsburgh Sleep Quality Index (PSQI) to assess perceived sleep quality reflective of the one-month period leading into the study. The global PSQI score can range from 0 to 21 points.
Urine electrolytes | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Researchers will analyze 24-hour urine samples for electrolytes (Na, K, Cl) content using the SmartLyte Electrolyte Analyzer. The unit of measure for Na, K, and Cl is milliequivalents (mEq).
Inflammatory cytokine responses | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Plasma will be used for a multiplex to measure inflammatory cytokines tumor necrosis factor-alpha, interleukin-6, monocyte chemoattractant protein-1, and interleukin-1. These biomarkers will be measured by enzyme-linked immunosorbent assays (ELISAs) from R&D.
Dietary intake | Change score from habitual consumption to after the hydration interventions (2 weeks)
  The investigators will instruct participants to complete a diet log for 3 days which will be operationalized with Nutrition Data System for Research (NDSR).

OTHER OUTCOMES:
Hemoglobin | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Whole blood samples will be analyzed for hemoglobin concentration (HemoCue, radiometer)
Hematocrit | Change score from habitual consumption to after the hydration interventions (2 weeks)
  Whole blood samples will be analyzed for hematocrit as a percentage (Thermo Hematocrit Microcentrifuge).
Physical activity | Pre-intervention (intake visit)
  Participants will wear an ActiGraph GT3X accelerometer for 14 days to objectively quantify steps taken per day.
Area deprivation index | Pre-intervention (intake visit)
  Investigators will measure participant's area deprivation index (ADI) based on their self-reported zip code. The ADI is a multidimensional assessment of a region's socioeconomic conditions. It is used to measure and quantify the level of deprivation or disadvantage experienced by residents in a specific geographical area. The composite score will be standardized to have a mean of 100 and a standard deviation of 20 to assist interpretation.
Blood pressure reactivity responses | Change score from habitual consumption to after the hydration interventions (2 weeks)
  The investigators will measure systolic and diastolic pressure using photoplethysmography at the finger and manually measure brachial pressures in millimeters of mercury. Systolic and diastolic blood pressure will be assessed at rest and during a cold pressor test. Blood pressure reactivity will be expressed as a change in pressure (mmHg) from baseline to the last 30 seconds of the cold pressor test.

CONTACTS AND LOCATIONS:
Overall Officials: Austin T Robinson, Ph.D., Study Director — Indiana University; L. Bruce Gladden, Ph.D., Study Director — Auburn University
Locations (1):
- Kinesiology Building, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Unidentified individual participant data will be made available to other researchers upon reasonable request and data and material transfer agreement
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years after completion of the study, indefinitely
Access Criteria: Unidentified individual participant data will be made available to other researchers upon reasonable request and data and completion of a material transfer agreement with Auburn University.

REFERENCES:
- [Background] Robinson AT, Linder BA, Barnett AM, Jeong S, Sanchez SO, Nichols OI, McIntosh MC, Hutchison ZJ, Tharpe MA, Watso JC, Gutierrez OM, Fuller-Rowell TE. Cross-sectional analysis of racial differences in hydration and neighborhood deprivation in young adults. Am J Clin Nutr. 2023 Oct;118(4):822-833. doi: 10.1016/j.ajcnut.2023.08.005. Epub 2023 Aug 22. PMID 37619651
- [Background] Fuller-Rowell TE, Nichols OI, Robinson AT, Boylan JM, Chae DH, El-Sheikh M. Racial disparities in sleep health between Black and White young adults: The role of neighborhood safety in childhood. Sleep Med. 2021 May;81:341-349. doi: 10.1016/j.sleep.2021.03.007. Epub 2021 Mar 12. PMID 33798979
- [Background] Brooks CJ, Gortmaker SL, Long MW, Cradock AL, Kenney EL. Racial/Ethnic and Socioeconomic Disparities in Hydration Status Among US Adults and the Role of Tap Water and Other Beverage Intake. Am J Public Health. 2017 Sep;107(9):1387-1394. doi: 10.2105/AJPH.2017.303923. Epub 2017 Jul 20. PMID 28727528
- [Background] Onufrak SJ, Park S, Sharkey JR, Sherry B. The relationship of perceptions of tap water safety with intake of sugar-sweetened beverages and plain water among US adults. Public Health Nutr. 2014 Jan;17(1):179-85. doi: 10.1017/S1368980012004600. Epub 2012 Oct 26. PMID 23098620
- [Background] Onufrak SJ, Park S, Sharkey JR, Merlo C, Dean WR, Sherry B. Perceptions of tap water and school water fountains and association with intake of plain water and sugar-sweetened beverages. J Sch Health. 2014 Mar;84(3):195-204. doi: 10.1111/josh.12138. PMID 24443781
- [Background] Park S, Onufrak SJ, Cradock AL, Patel A, Hecht C, Blanck HM. Perceptions of Water Safety and Tap Water Taste and Their Associations With Beverage Intake Among U.S. Adults. Am J Health Promot. 2023 Jun;37(5):625-637. doi: 10.1177/08901171221150093. Epub 2023 Jan 6. PMID 36609168